CLINICAL TRIAL: NCT04718259
Title: Evaluation of the Intraoperative and PO Analgesic Outcome of Using Midazolam as Adjuvant to Bupivacaine Intrathecal Anesthesia for Children Undergoing Lower Abdominal Surgeries.
Brief Title: The Use of Midazolam as Adjuvant to Bupivacaine Intrathecal Anesthesia for Children Undergoing Lower Abdominal Surgeries.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, MOHAMMED FAWZI ALI ABOSAMAK, consultant anesthesia, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: Intrathecal midazolam
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Analgesia; Children, Only; Bupivacaine; Midazolam
MeSH Terms: conditions — Agnosia | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Will include patients who will receive bupivacaine intrathecal injection without adjuvant.
  Interventions: Drug: intrathecal bupivacaine
- Group B (Experimental): Will include patients who will receive bupivacaine and midazolam.
  Interventions: Drug: intrathecal bupivacaine; Drug: midazolam

INTERVENTIONS:
Drug: intrathecal bupivacaine — The use of intrathecal bupivacaine will be compared to the use of intrathecal bupivacaine and midazolam.
  Other Names: intrathecal bupivacaine and midazolam
Drug: midazolam — midazolam
  Arms: Group B

SUMMARY:
The study will be carried on children undergoing lower abdominal surgeries. Patients will be randomly categorized into two study groups. Group A will include patients who will receive bupivacaine intrathecal injection without adjuvant. Group B will include patients who will receive bupivacaine and preservative-free midazolam.

ELIGIBILITY:
Inclusion Criteria:

* All children aged 3-12 years, assigned for lower abdominal and pelvic surgeries and will be ASA grade I after obtaining written fully informed parental consent.

Exclusion Criteria:

* Patients with congenital anomalies especially of the spine, infections in the skin of the back, had coagulopathy, or allergy to the study drugs and those whose parents refused to give the consent .

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2020-01-18 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative analgesia | 90 days
  Efficacy of PO analgesia will be determined, by an assistant who will be blinded about the using the observational pain-discomfort scale (OPS), which assesses behavioral parameters that can be evaluated objectively.
Duration of analgesia | 90 days
  defined as the time elapsed since end of the surgical procedure till OPS reaches >11
Post operative resolution of motor block | 90 days
  will be assessed using Bromage score till complete recovery.
The level of Post operative sedation | 90 days
  will be assessed at 30 & 120 minutes after admission to the recovery room using the modified WilsonSedation Score (WSS)
PO hospital stay | 90 days
  Duration of PO hospital stay

SECONDARY OUTCOMES:
The rate of procedural success | 90 days
  Defined as peak sensory level at least T10, Bromage score at 3 at 10-min after spina block and no response to surgical stimuli once surgery will be allowed to start.

CONTACTS AND LOCATIONS:
Locations (1):
- Alemeis hospital ksa, Jizan, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided
After analyzing the data.